CLINICAL TRIAL: NCT02110602
Title: Short-term Dietary Intake and Branched Chain Amino Acids
Brief Title: Dietary Intake and Circulating Levels of Branched Chain Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Geoffrey Walford, MD, Geoffrey Walford, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013P002607
Record Dates: First submitted 2014-03-12; First posted 2014-04-10 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Dietary Intake of Branched Chain Amino Acids
Keywords: Nutrition
MeSH Terms: interventions — Isoleucine; Leucine; Valine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial Diet - high in amino acid levels (Experimental): Visit 1 (Day 1): Screening Visit
  Visit 2 (14-21 days after Visit 1): Begin high amino acid diet
  Visit 3 (4 days after Visit 2): Completion of high amino acid diet
  Visit 4 (3 days after Visit 3): Begin low amino acid diet
  Visit 5 (4 days after Visit 4): Completion of low amino acid diet, completion of study
  Interventions: Other: Diet high in amino acid levels; Other: Diet low in amino acid levels
- Initial Diet - low in amino acid levels (Experimental): Visit 1 (Day 1): Screening Visit
  Visit 2 (14-21 days after Visit 1): Begin low amino acid diet
  Visit 3 (4 days after Visit 2): Completion of low amino acid diet
  Visit 4 (3 days after Visit 3): Begin high amino acid diet
  Visit 5 (4 days after Visit 4): Completion of high amino acid diet, completion of study
  Interventions: Other: Diet high in amino acid levels; Other: Diet low in amino acid levels

INTERVENTIONS:
Other: Diet high in amino acid levels — Meals will be prepared in the Clinical Research Center Metabolism & Nutrition Metabolic Kitchen, and participants will eat only this food during the controlled-diet periods of the study. The diets will contain equivalent calories (matched to the requirements of each participant) and either a low or high percentage of all BCAAs relative to protein content.
  Other Names: Amino Acid supplements to be used in prepared meals:; Vitaflo MSUD express; l-isoleucine; l-leucine; l-valine
Other: Diet low in amino acid levels — Meals will be prepared in the Clinical Research Center Metabolism & Nutrition Metabolic Kitchen, and participants will eat only this food during the controlled-diet periods of the study. The diets will contain equivalent calories (matched to the requirements of each participant) and either a low or high percentage of all BCAAs relative to protein content.

SUMMARY:
The investigators are conducting this research study to find out if eating low or high levels of specific amino acids changes the levels of these same amino acids in the blood. Amino acids are the building blocks of protein that are normally found in food. The amino acids the investigators are studying are called branched chain amino acids. The investigators will look at the levels (amount) of branched chain amino acids in blood before and after consumption of specially prepared meals. The investigators hypothesize that circulating branch chain amino acid (BCAA) levels will be lower following a low BCAA-content diet compared with a high BCAA-content diet.

ELIGIBILITY:
Inclusion Criteria:

* Adult males
* Ages 20-40
* Healthy

Exclusion Criteria:

* Age less than 20 or greater than 40
* Female sex
* Use of medications and herbal or vitamin supplements during the study or less than one month prior to enrollment in the study
* Body mass index (BMI) less than 20 or greater than 25
* Changes of more than 5 pounds in weight (increase or decrease) during the month prior to enrollment in the study
* Participation in more than 300 minutes of exercise per week during the month prior to enrollment in the study or plans for changes in exercise level during the study
* Known diabetes or pre-diabetes (based on prior diagnoses; use of medications to lower glucose; or fasting blood glucose > 100mg/dL at screening)
* Untreated hypertension (defined as systolic blood pressure > 140mmHg and diastolic blood pressure > 90mmHg)
* Use of nicotine-containing products, including those inhaled, chewed, or patches during the study.
* Use of drugs of abuse.
* Conditions causing intestinal malabsorption, including celiac disease or a history of intestinal or gastric surgery
* Restrictions that prevent adherence to standardized meals or unwillingness to adhere to a pre-specified meal plan, including abstinence from alcohol and limitation to 1 caffeinated beverage per day
* Known anemia (men, hematocrit < 38%) based on prior testing

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Comparison of Branch Chain Amino Acid levels following diet interventions | 4 days
  A comparison of branched chain amino acid levels (as measured by mass spectrometry) following 4 days of a low and following 4 days of a high BCAA-content diet

SECONDARY OUTCOMES:
Change in fasting BCAA levels from native dietary intake to completion of diet intervention | 4 days

OTHER OUTCOMES:
Comparison of fasting glucose and insulin levels following diet interventions | 4 days
Change in fasting glucose and insulin levels from native dietary intake to completion of diet intervention | 4 days
Tolerance of diet interventions | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Walford, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Cavallaro NL, Garry J, Shi X, Gerszten RE, Anderson EJ, Walford GA. A pilot, short-term dietary manipulation of branched chain amino acids has modest influence on fasting levels of branched chain amino acids. Food Nutr Res. 2016 Jan 14;60:28592. doi: 10.3402/fnr.v60.28592. eCollection 2016. PMID 26781817